CLINICAL TRIAL: NCT01641614
Title: Clinical and Ultramicroscopic Myocardial Randomized Study of On-Pump Beating Heart Mitral Valve Replacement
Brief Title: Beating Versus Arrested Heart for Mitral Valve Replacement
Acronym: BAHMVR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Clotario Neptali Carrasco Cueva, Medical Doctor , Profesor of Cardiac Surgery, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REQ:690
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Mitral Stenosis; Mitral Insufficiency
Keywords: Mitral valve; valve replacement; arrested heart; beating heart
MeSH Terms: conditions — Mitral Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beating heart surgery (Experimental): Group A (Beating heart) surgery was performed under normal temperature (36⁰ C) ,once CPB was established, the patient was placed in Trendelenburg position and a retrograde perfusion catheter was inserted into the coronary sinus and ligated by a simple suture line. Aorta cross clamping was immediately established and blood was oxygenated and delivered continuously through a catheter Mitral valve was exposed using the left atrial retractor. Mitral valve replacement (MVR) was performed using a metallic or bioprostheses substitution by interrupted suture De Vegas' technique.
  Interventions: Procedure: Mitral valve replacement
- heart surgery Group B (Active Comparator): Group B (arrested heart) surgery was performed under moderate hypothermia (32⁰C) as technique requirement (3). After cardiac arrest, during the period of cross clamping, the aortic root was perfused through the cardioplegias's cannula with oxygenated blood at a rate between 200 mL/min to 300 mL/min for 2 minutes with 15 minutes intervals.Mitral valve replacement (MVR) was performed using a metallic or bioprostheses substitution by interrupted suture De Vegas' technique.
  Interventions: Procedure: mitral valve replacement

INTERVENTIONS:
Procedure: Mitral valve replacement — Mitral valve replacement (MVR) was performed using a metallic or bioprostheses substitution by interrupted suture. For the beating heart the prostheses was functionally tested before removal of the retrograde perfusion catheter and for the arrested heart the prosthesis was artificially tested by pumping saline into the left ventricle. The tricuspid valve repair was done following De Vegas' technique in both groups
  Arms: Beating heart surgery
Procedure: mitral valve replacement — Mitral valve replacement (MVR) was performed using a metallic or bioprostheses substitution by interrupted suture. For the beating heart the prostheses was functionally tested before removal of the retrograde perfusion catheter and for the arrested heart the prosthesis was artificially tested by pumping saline into the left ventricle. The tricuspid valve repair was done following De Vegas' technique in both groups
  Arms: heart surgery Group B

SUMMARY:
The purpose of this study is to evaluate the immediately clinic and ultramicroscopic myocardial cellular ischemia and reperfusion to replace of the mitral valve using arrested heart versus on-pump empty beating heart surgical techniques.

DETAILED DESCRIPTION:
During open-heart surgery prevention of ischemia and reperfusion following cardioplegic arrest are essential for myocardial protection. Beating heart surgery on normothermic bypass simulates physiologic cardiac status and is good method for myocardial protection. A comparison of both available techniques for valve replacement arrested heart versus on-pump empty beating heart of the clinical and ultramicroscopic myocardial alterations will allowed to better understand myocardial protection because eliminated the use of cardioplegia and the corollary risk of ischemic reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* all patient included into the study were adults 18-60 years old,
* with an echocardiography diagnosis of mitral and/or tricuspid valve disease due to inflammatory acquired diseases,
* no previous history of cardiac surgery and d) elective indication for valve replacement.

Exclusion Criteria:

* with metabolic diseases such as diabetes mellitus and uremia,
* with coronary artery diseases,
* dilated myocardiopathy,
* with severe chronic pulmonary obstructive diseases,
* with present or past history of malignant diseases,
* acute endocarditis
* with severe pre-operatory laboratory parameters such as creatinine levels > 3mg/dL, Hemoglobin ≤ 7.0 g/dL, Prothrombin time/activity ≤ 70% and clotting time ≥ 10 minutes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
mitral valve replacement | 1hour , 3 hours and 1 hour after surgery procedure
  Mitral valve replacement (MVR) was performed using a metallic or bioprostheses substitution by interrupted suture. For the beating heart the prostheses was functionally tested before removal of the retrograde perfusion catheter and for the arrested heart the prosthesis was artificially tested by pumping saline into the left ventricle. The tricuspid valve repair was done following De Vegas' technique in both groups with the beating heart also in the group B.

SECONDARY OUTCOMES:
Ultramicroscopic evidences of ischemia | 1hour, 3 hours and 1 hour after aortic clamping
  During the surgery myocardial biopsies were performed as full thickness transmural specimen of three small fragments for electromicrospic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ana Neri, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] Schaper J, Schwarz F, Kittstein H, Stammler G, Winkler B, Scheld H, Hehrlein F. The effects of global ischemia and reperfusion on human myocardium: quantitative evaluation by electron microscopic morphometry. Ann Thorac Surg. 1982 Feb;33(2):116-22. doi: 10.1016/s0003-4975(10)61895-4. PMID 7065773
- [Background] Babaroglu S, Yay K, Parlar AI, Ates C, Mungan U, Cicekcioglu F, Tutun U, Katircioglu SF. Beating heart versus conventional mitral valve surgery. Interact Cardiovasc Thorac Surg. 2011 Mar;12(3):441-7. doi: 10.1510/icvts.2010.255240. Epub 2010 Dec 21. PMID 21177299
- [Background] Kaplon RJ, Pham SM, Salerno TA. Beating-heart valvular surgery: a possible alternative for patients with severely compromised ventricular function. J Card Surg. 2002 Mar-Apr;17(2):170-2. doi: 10.1111/j.1540-8191.2002.tb01194.x. PMID 12220071
- [Background] Matsumoto Y, Watanabe G, Endo M, Sasaki H, Kasashima F, Kosugi I. Efficacy and safety of on-pump beating heart surgery for valvular disease. Ann Thorac Surg. 2002 Sep;74(3):678-83. doi: 10.1016/s0003-4975(02)03753-0. PMID 12238823
- [Background] Salhiyyah K, Taggart D. Beating-heart valve surgery: A systematic review. Asian Cardiovasc Thorac Ann. 2009 Dec;17(6):650-8. doi: 10.1177/0218492309348942. PMID 20026547
- [Background] Ghosh S, Jutley RS, Wraighte P, Shajar M, Naik SK. Beating-heart mitral valve surgery in patients with poor left ventricular function. J Heart Valve Dis. 2004 Jul;13(4):622-7; discussion 627-9. PMID 15311869
- [Background] Mizuno T, Arai H. On-pump beating-heart mitral valve plasty without aortic cross-clamping. Jpn J Thorac Cardiovasc Surg. 2006 Oct;54(10):454-7. doi: 10.1007/s11748-006-0031-4. PMID 17087329
- [Background] Bara C, Zhang R, Haverich A. De Vega annuloplasty for tricuspid valve repair in posttraumatic tricuspid insufficiency--16 years experience. Int J Cardiol. 2008 Jun 6;126(3):e61-2. doi: 10.1016/j.ijcard.2007.01.027. Epub 2007 Mar 29. PMID 17395296
- [Background] Hassan HT, Veit A, Maurer HR. Synergistic interactions between differentiation-inducing agents in inhibiting the proliferation of HL-60 human myeloid leukaemia cells in clonogenic micro assays. J Cancer Res Clin Oncol. 1991;117(3):227-31. doi: 10.1007/BF01625429. PMID 1709642
- [Background] Herrera JM, Cuenca J, Campos V, Rodriguez F, Vicente Valle J, Juffe A. [Coronary surgery without extracorporeal circulation: 5-year experience]. Rev Esp Cardiol. 1998 Feb;51(2):136-40. Spanish. PMID 9542436
- [Background] Karolak W, Hirsch G, Buth K, Legare JF. Medium-term outcomes of coronary artery bypass graft surgery on pump versus off pump: results from a randomized controlled trial. Am Heart J. 2007 Apr;153(4):689-95. doi: 10.1016/j.ahj.2007.01.033. PMID 17383313
- [Background] Karadeniz U, Erdemli O, Yamak B, Genel N, Tutun U, Aksoyek A, Cicekcioglu F, Parlar AI, Katircioglu SF. On-pump beating heart versus hypothermic arrested heart valve replacement surgery. J Card Surg. 2008 Mar-Apr;23(2):107-13. doi: 10.1111/j.1540-8191.2007.00536.x. PMID 18304123
- [Background] Lichtenstein SV, Ashe KA, el Dalati H, Cusimano RJ, Panos A, Slutsky AS. Warm heart surgery. J Thorac Cardiovasc Surg. 1991 Feb;101(2):269-74. PMID 1992237
- [Background] Kamlot A, Bellows SD, Simkhovich BZ, Hale SL, Aoki A, Kloner RA, Kay GL. Is warm retrograde blood cardioplegia better than cold for myocardial protection? Ann Thorac Surg. 1997 Jan;63(1):98-104. doi: 10.1016/s0003-4975(96)01074-0. PMID 8993249
- [Background] Eke CC, Gundry SR, Fukushima N, Bailey LL. Is there a safe limit to coronary sinus pressure during retrograde cardioplegia? Am Surg. 1997 May;63(5):417-20. PMID 9128230
- [Background] Gundry SR, Wang N, Sciolaro CM, Van Arsdell GS, Razzouk AJ, Hill AC, Bailey LL. Uniformity of perfusion in all regions of the human heart by warm continuous retrograde cardioplegia. Ann Thorac Surg. 1996 Jan;61(1):33-5. doi: 10.1016/0003-4975(95)00880-2. PMID 8561599
- [Background] Pena E, Solano L, Portillo Z, Meertens de Rodriguez L. [Nutritional status of institutionalized elderly. Valencia, State of Carabobo, Venezuela]. Arch Latinoam Nutr. 1998 Jun;48(2):104-11. Spanish. PMID 9830484